CLINICAL TRIAL: NCT07233915
Title: Genetic Profile in Patients With Ruptured and Unruptured Intracranial Aneurysms: Observational Study Aimed at Identifying Genetic Variants Associated With the Risk of Intracranial Aneurysm Rupture
Brief Title: Genetic Profile In Patients With Ruptured and Unruptured Intracranial Aneurysms
Acronym: ANEUBIO
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: ANEUBIO
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Aneurism
Keywords: Rupture risk; Genetic factors; Observational study; Biobank; Intracranial aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project will involve multiple units within our Institute (Neurosurgery, Cerebrovascular Diseases, Neurology IV), as well as additional neurosurgical centers across Italy, for the enrollment of patients with saccular intracranial aneurysms (sIA), both ruptured and unruptured. Based on predefined inclusion and exclusion criteria, the recruitment target over a two-year period is 400 patients with sIA (200 ruptured, 200 unruptured) and 200 healthy controls. The study will not alter clinical practice: treatment decisions for unruptured sIA will be made independently by vascular teams according to routine standards.

For each enrolled subject, anonymized clinical data will be collected (age, sex, BMI, lifestyle habits, family history, comorbidities, aneurysmal parameters) to build an integrated database within the Biorepository. Peripheral blood samples will be obtained for genomic analyses, and when available (e.g., during clipping procedures or lumbar puncture), aneurysm wall tissue and/or cerebrospinal fluid (CSF) samples will be collected for expression studies. All materials and data (clinical/genetic) will be coded and stored at the Cryobank of the Fondazione IRCCS Istituto Neurologico Besta.

Genomic analyses: a pathway-based Genome-Wide Association Study (GWAS) is planned.

Phase I: Genotyping of 200 patients (100 with ruptured sIA, 100 with unruptured sIA) and 100 healthy controls, with combined analysis of genetic data and environmental factors related to rupture risk.

Phase II: Validation in an additional cohort of 200 patients (100 ruptured, 100 unruptured) and 100 controls to confirm the associations of identified SNPs.

DETAILED DESCRIPTION:
This observational study aims to identify potential genetic determinants associated with the risk of rupture in saccular intracranial aneurysms (sIA). The study is conducted in collaboration with three Units of the Fondazione IRCCS Istituto Neurologico Carlo Besta in Milan (Neurosurgery Unit II, Cerebrovascular Diseases Unit, Neurology Unit IV), as well as additional neurosurgical centers across Italy, particularly for the enrollment of patients with ruptured sIA who do not present to Besta due to the absence of an Emergency Department.

As an observational study, it does not involve any modification to the routine clinical management of patients with sIA at participating centers. Specifically, the decision to propose surgical or endovascular treatment for patients with ruptured or unruptured aneurysms will be made independently of the study, based on shared criteria discussed during regular multidisciplinary vascular meetings. Furthermore, no additional follow-up is planned beyond what is routinely scheduled for patients undergoing surgical or endovascular treatment for intracranial aneurysms.

Each patient will be asked to provide informed consent through a dedicated form. Once consent is obtained, each participant will be assigned a unique alphanumeric central code, used exclusively for study purposes. Throughout the duration of the project and thereafter, only the responsible physician will be able to link the code to the patient's identity.

Patients will undergo clinical evaluation at the time of enrollment, as part of standard clinical practice. Anonymized clinical data will be recorded in a centralized database and will include: sex, age, height, weight, regular use of illicit substances, alcohol consumption, smoking habits, family history of sIA, arterial hypertension, medical history with particular attention to autoimmune diseases and recent infections, general and neurological assessment, and aneurysmal characteristics (location, maximum diameter, morphology-regular or irregular).

Each patient will also undergo peripheral venous blood sampling for genomic studies. When available (e.g., during clipping procedures or lumbar puncture performed for decompression or other clinical indications), samples of aneurysm wall tissue, subcutaneous arterial wall, and/or cerebrospinal fluid (CSF) will be collected. Biological samples, along with coded clinical and genetic data, will be stored at the Fondazione IRCCS Istituto Neurologico Carlo Besta in separate containers, housed in controlled and locked environments, to establish the first Integrated Italian Biobank for Intracranial Aneurysms.

Regarding genomic analyses, a pathway-based genome-wide association study (GWAS) will be conducted.

* Phase I: DNA extracted and genotyped from 200 patients (100 with ruptured sIA and 100 with unruptured sIA) and 100 healthy controls will be analyzed. Statistical analysis will assess the combined effect of genetic and environmental factors on rupture risk. In this phase, healthy subjects and patients with unruptured sIA will serve as control groups for patients with ruptured sIA.
* Phase II: An additional cohort of 200 patients (100 ruptured, 100 unruptured) and 100 healthy controls will be analyzed to validate the single nucleotide polymorphism (SNP) combinations identified in the preliminary phase.

Finally, the genetic and clinical data obtained from the biostatistical analysis of the entire cohort (400 patients and 200 healthy controls) will be used to develop a user-friendly computational tool aimed at estimating the individual risk of rupture in patients with sIA.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years, of both sexes
* Patients diagnosed with ruptured or unruptured saccular intracranial aneurysms (sIA)

Exclusion Criteria:

* Patients with non-saccular intracranial aneurysms
* Patients unable to provide informed consent due to language impairment or altered consciousness, in the absence of a legally appointed guardian

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ruptured or unruptured saccular intracranial aneurysms (sIA)
Sampling Method: Non-Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2014-02-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic variants | Within 2 years from patient enrollment and genotyping (Phase I and Phase II).
  Identification of genetic variants associated with the risk of rupture in patients with saccular intracranial aneurysms (sIA), through a pathway-based genome-wide association study (GWAS).

SECONDARY OUTCOMES:
Development of a tool to estimate Rupture Risk | Within 3 years, following completion of biostatistical analysis.
  Development of a user-friendly computational tool to estimate individual rupture risk in patients with unruptured sIA, based on combined genetic and clinical data.
Creation of a Biobank | Ongoing during the 2-year enrollment period and maintained beyond study completion.
  Creation of an integrated biobank including biological samples (aneurysm wall, CSF, control arterial wall), genetic profiles, and anonymized clinical data from patients with ruptured and unruptured sIA.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yasuno K, Bakircioglu M, Low SK, Bilguvar K, Gaal E, Ruigrok YM, Niemela M, Hata A, Bijlenga P, Kasuya H, Jaaskelainen JE, Krex D, Auburger G, Simon M, Krischek B, Ozturk AK, Mane S, Rinkel GJ, Steinmetz H, Hernesniemi J, Schaller K, Zembutsu H, Inoue I, Palotie A, Cambien F, Nakamura Y, Lifton RP, Gunel M. Common variant near the endothelin receptor type A (EDNRA) gene is associated with intracranial aneurysm risk. Proc Natl Acad Sci U S A. 2011 Dec 6;108(49):19707-12. doi: 10.1073/pnas.1117137108. Epub 2011 Nov 21. PMID 22106312
- [Background] Yasuno K, Bilguvar K, Bijlenga P, Low SK, Krischek B, Auburger G, Simon M, Krex D, Arlier Z, Nayak N, Ruigrok YM, Niemela M, Tajima A, von und zu Fraunberg M, Doczi T, Wirjatijasa F, Hata A, Blasco J, Oszvald A, Kasuya H, Zilani G, Schoch B, Singh P, Stuer C, Risselada R, Beck J, Sola T, Ricciardi F, Aromaa A, Illig T, Schreiber S, van Duijn CM, van den Berg LH, Perret C, Proust C, Roder C, Ozturk AK, Gaal E, Berg D, Geisen C, Friedrich CM, Summers P, Frangi AF, State MW, Wichmann HE, Breteler MM, Wijmenga C, Mane S, Peltonen L, Elio V, Sturkenboom MC, Lawford P, Byrne J, Macho J, Sandalcioglu EI, Meyer B, Raabe A, Steinmetz H, Rufenacht D, Jaaskelainen JE, Hernesniemi J, Rinkel GJ, Zembutsu H, Inoue I, Palotie A, Cambien F, Nakamura Y, Lifton RP, Gunel M. Genome-wide association study of intracranial aneurysm identifies three new risk loci. Nat Genet. 2010 May;42(5):420-5. doi: 10.1038/ng.563. Epub 2010 Apr 4. PMID 20364137
- [Background] Vlak MH, Algra A, Brandenburg R, Rinkel GJ. Prevalence of unruptured intracranial aneurysms, with emphasis on sex, age, comorbidity, country, and time period: a systematic review and meta-analysis. Lancet Neurol. 2011 Jul;10(7):626-36. doi: 10.1016/S1474-4422(11)70109-0. PMID 21641282
- [Background] Ruigrok YM, Rinkel GJ. Genetics of intracranial aneurysms. Stroke. 2008 Mar;39(3):1049-55. doi: 10.1161/STROKEAHA.107.497305. Epub 2008 Feb 7. PMID 18258833
- [Background] Liberzon A, Subramanian A, Pinchback R, Thorvaldsdottir H, Tamayo P, Mesirov JP. Molecular signatures database (MSigDB) 3.0. Bioinformatics. 2011 Jun 15;27(12):1739-40. doi: 10.1093/bioinformatics/btr260. Epub 2011 May 5. PMID 21546393
- [Background] Kurki MI, Hakkinen SK, Frosen J, Tulamo R, von und zu Fraunberg M, Wong G, Tromp G, Niemela M, Hernesniemi J, Jaaskelainen JE, Yla-Herttuala S. Upregulated signaling pathways in ruptured human saccular intracranial aneurysm wall: an emerging regulative role of Toll-like receptor signaling and nuclear factor-kappaB, hypoxia-inducible factor-1A, and ETS transcription factors. Neurosurgery. 2011 Jun;68(6):1667-75; discussion 1675-6. doi: 10.1227/NEU.0b013e318210f001. PMID 21336216
- [Background] Juvela S. Prehemorrhage risk factors for fatal intracranial aneurysm rupture. Stroke. 2003 Aug;34(8):1852-7. doi: 10.1161/01.STR.0000080380.56799.DD. Epub 2003 Jun 26. PMID 12829865
- [Background] Juvela S. Natural history of unruptured intracranial aneurysms: risks for aneurysm formation, growth, and rupture. Acta Neurochir Suppl. 2002;82:27-30. doi: 10.1007/978-3-7091-6736-6_5. PMID 12378985
- [Background] Johnston SC, Selvin S, Gress DR. The burden, trends, and demographics of mortality from subarachnoid hemorrhage. Neurology. 1998 May;50(5):1413-8. doi: 10.1212/wnl.50.5.1413. PMID 9595997
- [Background] Hahn LW, Ritchie MD, Moore JH. Multifactor dimensionality reduction software for detecting gene-gene and gene-environment interactions. Bioinformatics. 2003 Feb 12;19(3):376-82. doi: 10.1093/bioinformatics/btf869. PMID 12584123
- [Background] Frosen J, Piippo A, Paetau A, Kangasniemi M, Niemela M, Hernesniemi J, Jaaskelainen J. Remodeling of saccular cerebral artery aneurysm wall is associated with rupture: histological analysis of 24 unruptured and 42 ruptured cases. Stroke. 2004 Oct;35(10):2287-93. doi: 10.1161/01.STR.0000140636.30204.da. Epub 2004 Aug 19. PMID 15322297
- [Background] de Rooij NK, Linn FH, van der Plas JA, Algra A, Rinkel GJ. Incidence of subarachnoid haemorrhage: a systematic review with emphasis on region, age, gender and time trends. J Neurol Neurosurg Psychiatry. 2007 Dec;78(12):1365-72. doi: 10.1136/jnnp.2007.117655. Epub 2007 Apr 30. PMID 17470467
- [Background] Bilguvar K, Yasuno K, Niemela M, Ruigrok YM, von Und Zu Fraunberg M, van Duijn CM, van den Berg LH, Mane S, Mason CE, Choi M, Gaal E, Bayri Y, Kolb L, Arlier Z, Ravuri S, Ronkainen A, Tajima A, Laakso A, Hata A, Kasuya H, Koivisto T, Rinne J, Ohman J, Breteler MM, Wijmenga C, State MW, Rinkel GJ, Hernesniemi J, Jaaskelainen JE, Palotie A, Inoue I, Lifton RP, Gunel M. Susceptibility loci for intracranial aneurysm in European and Japanese populations. Nat Genet. 2008 Dec;40(12):1472-7. doi: 10.1038/ng.240. Epub 2008 Nov 9. PMID 18997786
- [Background] Barrett JC, Fry B, Maller J, Daly MJ. Haploview: analysis and visualization of LD and haplotype maps. Bioinformatics. 2005 Jan 15;21(2):263-5. doi: 10.1093/bioinformatics/bth457. Epub 2004 Aug 5. PMID 15297300